CLINICAL TRIAL: NCT00862849
Title: Phase 1, Randomized, Double-Blind, Pharmacokinetic and Glucodynamic 6-Way Crossover Study of SC Administered Insulin Lispro With Recombinant Human Hyaluronidase (rHuPH20) and Regular Human Insulin With Recombinant Human Hyaluronidase (rHuPH20) Compared to Insulin Lispro Alone in Healthy Volunteers
Brief Title: Pharmacokinetic and Glucodynamic Crossover Study of Subcutaneously (SC) Administered Insulin Lispro + Recombinant Human Hyaluronidase (rHuPH20) and Regular Human Insulin + rHuPH20 Compared to Insulin Lispro Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Double
Other Study IDs: HALO-117-103
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus
Keywords: rHuPH20; Recombinant Human Hyaluronidase; Insulin Lispro; Regular Human Insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Lispro; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin Lispro, Regular Human Insulin, rHuPH20 (Experimental): All participants were randomized to 1 of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, or CBA), each of which was comprised of the same 3 interventions (A, B, and C).
  Intervention A: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) insulin lispro with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Intervention B: a single, SC injection of 0.15 U/kg regular human insulin (RHI) with 3.75 ng/kg rHuPH20
  Intervention C: a single, SC injection of 0.15 U/kg insulin lispro alone
  There was a washout period of 3 to 14 days between interventions.
  The treatment sequence (ABC, ACB, BAC, BCA, CAB, or CBA) was repeated once so that each participant received up to 6 injections.
  Interventions: Drug: Insulin Lispro; Drug: Regular Human Insulin; Drug: rHuPH20

INTERVENTIONS:
Drug: Insulin Lispro
  Other Names: Humalog
Drug: Regular Human Insulin
  Other Names: RHI; Humulin R
Drug: rHuPH20
  Other Names: recombinant human hyaluronidase; HYLENEX

SUMMARY:
Insulin lispro and regular human insulin are Food and Drug Administration (FDA)-approved medications for the treatment of diabetes mellitus. Recombinant human hyaluronidase (rHuPH20) is approved by the FDA as an aid to the absorption and dispersion of other injectable drugs. In this study, rHuPH20 will be co-administered with both insulin lispro and regular human insulin in order to determine if it improves the absorption of these insulins to more closely mimic the body's natural increase in insulin in response to a meal.

DETAILED DESCRIPTION:
The purpose of this study is to compare the pharmacokinetics (absorption, distribution, breakdown and elimination) of regular human insulin + recombinant human hyaluronidase (rHuPH20) versus insulin lispro alone, and to compare the pharmacokinetics of insulin lispro + rHuPH20 versus insulin lispro alone. The effects of regular human insulin + rHuPH20, insulin lispro + rHuPH20, and insulin lispro alone on the body will be evaluated by blood glucose measurements and by calculating the rate at which a glucose solution is infused to maintain blood glucose within a certain range. The safety and tolerability of insulin lispro with and without rHuPH20 and regular human insulin with rHuPH20 will be studied. The study drugs will be administered by subcutaneous (under the skin) injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities.)
* Body mass index (BMI) between 18-27 kilograms per meter squared (kg/m^2), inclusive.
* Total body weight >65 kilograms (kg) (143 pounds [lb]) for men and >46 kg (101 lb) for women.
* Decision making capacity and willingness to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including adequate venous access.
* Vital signs (blood pressure, pulse rate, body temperature) within normal range or, if out of range, assessed by the Principal Investigator (PI) as not clinically significant (NCS).
* Fasting blood glucose level <100 milligrams per deciliter (mg/dL) at screening.
* A negative serum pregnancy test (if female of childbearing potential).
* Female participants of childbearing potential must agree to be practicing effective birth control or abstinence currently and agree to continue to do so for the duration of their time on study.
* Signed, written Institutional Review Board (IRB)-approved informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, oncologic, or neurologic (to include history of seizures) disease; hypoglycemic episodes; intercurrent illness (such as influenza); or allergic disease (including severe drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). Clinical significance to be determined by the PI.
* As judged by the Investigator, clinically significant findings in routine laboratory data. (Anemia with hematocrit less than 33% at screening is specifically exclusionary.)
* Known history of diabetes mellitus (type 1 or type 2) or gestational diabetes.
* Known allergy to hyaluronidase or any other ingredient in the study drug.
* Positive human immunodeficiency virus (HIV 1) antibody test, hepatitis B (anti-hepatitis B surface antigen [anti-HBsAg]) or hepatitis C (anti-hepatitis C virus [anti-HCV]) antibody test.
* History or evidence of alcohol or drug abuse.
* History or evidence of use of any tobacco or nicotine-containing product within 6 months of screening and a screening qualitative urine nicotine test.
* Use of drugs that may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action or glucose utilization.
* Donation of blood in excess of 500 milliliters (mL) within 56 days before dosing.
* Participation in a study of any investigational drug or device 30 days before enrollment in this study.
* The participant is unfit for the study in the opinion of the Investigator.
* Women who are pregnant or breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Morrow, M.D., Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States

REFERENCES:
- [Result] Morrow L, Muchmore DB, Ludington EA, Vaughn DE, Hompesch M. Reduction in intrasubject variability in the pharmacokinetic response to insulin after subcutaneous co-administration with recombinant human hyaluronidase in healthy volunteers. Diabetes Technol Ther. 2011 Oct;13(10):1039-45. doi: 10.1089/dia.2011.0115. Epub 2011 Jun 29. PMID 21714645

RESULTS

PARTICIPANT FLOW:
Groups:
- Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone: Interventions 1 and 4: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) insulin lispro with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Interventions 2 and 5: a single, SC injection of 0.15 U/kg regular human insulin (RHI) with 3.75 ng/kg rHuPH20
  Interventions 3 and 6: a single, SC injection of 0.15 U/kg insulin lispro alone
  There was a washout period of 3 to 14 days between interventions. The sequence of interventions was repeated so that each participant received up to 6 injections.
- Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20: Interventions 1 and 4: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) insulin lispro with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Interventions 2 and 5: a single, SC injection of 0.15 U/kg insulin lispro alone
  Interventions 3 and 6: a single, SC injection of 0.15 U/kg regular human insulin (RHI) with 3.75 ng/kg rHuPH20
  There was a washout period of 3 to 14 days between interventions. The sequence of interventions was repeated so that each participant received up to 6 injections.
- RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone: Interventions 1 and 4: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) regular human insulin (RHI) with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Interventions 2 and 5: a single, SC injection of 0.15 U/kg insulin lispro with 3.75 ng/kg rHuPH20
  Interventions 3 and 6: a single, SC injection of 0.15 U/kg insulin lispro alone
  There was a washout period of 3 to 14 days between interventions. The sequence of interventions was repeated so that each participant received up to 6 injections.
- RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20: Interventions 1 and 4: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) regular human insulin (RHI) with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Interventions 2 and 5: a single, SC injection of 0.15 U/kg insulin lispro alone
  Interventions 3 and 6: a single, SC injection of 0.15 U/kg insulin lispro with 3.75 ng/kg rHuPH20
  There was a washout period of 3 to 14 days between interventions. The sequence of interventions was repeated so that each participant received up to 6 injections.
- Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20: Interventions 1 and 4: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) insulin lispro alone
  Interventions 2 and 5: a single, SC injection of 0.15 U/kg insulin lispro with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Interventions 3 and 6: a single, SC injection of 0.15 U/kg regular human insulin (RHI) with 3.75 ng/kg rHuPH20
  There was a washout period of 3 to 14 days between interventions. The sequence of interventions was repeated so that each participant received up to 6 injections.
- Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20: Interventions 1 and 4: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) insulin lispro alone
  Interventions 2 and 5: a single, SC injection of 0.15 U/kg regular human insulin (RHI) with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Interventions 3 and 6: a single, SC injection of 0.15 U/kg insulin lispro with 3.75 ng/kg rHuPH20
  There was a washout period of 3 to 14 days between interventions. The sequence of interventions was repeated so that each participant received up to 6 injections.
Period: Intervention 1
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 5 | 3 | 4 | 4 | 3
Received at Least One Dose of Study Drug | 3 | 5 | 3 | 4 | 4 | 3
Completed | 3 | 5 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1 (3 to 14 Days)
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 5 | 3 | 4 | 4 | 3
Completed | 3 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Intervention 2
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 4 | 3 | 4 | 4 | 3
Completed | 3 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2 (3 to 14 Days)
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 4 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Period: Intervention 3
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 3 (3 to 14 Days)
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 4
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 4 (3 to 14 Days)
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 5
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 5 (3 to 14 Days)
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 6
Arm/Group | Lispro+rHuPH20 First, Then RHI+rHuPH20, Then Lispro Alone | Lispro+rHuPH20 First, Then Lispro Alone, Then RHI+rHuPH20 | RHI+rHuPH20 First, Then Lispro+rHuPH20, Then Lispro Alone | RHI+rHuPH20 First, Then Lispro Alone, Then Lispro+rHuPH20 | Lispro Alone First, Then Lispro+rHuPH20, Then RHI+rHuPH20 | Lispro Alone First, Then RHI+rHuPH20, Then Lispro+rHuPH20
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of insulin lispro, regular human insulin, or recombinant human hyaluronidase (rHuPH20).
Groups:
- All Participants: All participants were randomized to 1 of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, or CBA), each of which was comprised of the same 3 interventions (A, B, and C).
  Intervention A: a single, subcutaneous (SC) injection of 0.15 units per kilogram (U/kg) insulin lispro with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20)
  Intervention B: a single, SC injection of 0.15 U/kg regular human insulin (RHI) with 3.75 ng/kg rHuPH20
  Intervention C: a single, SC injection of 0.15 U/kg insulin lispro alone
  There was a washout period of 3 to 14 days between interventions.
  The treatment sequence (ABC, ACB, BAC, BCA, CAB, or CBA) was repeated once so that each participant received up to 6 injections.
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Intra-participant Variability in Percent of Total Area Under the Plasma Insulin Concentration-Versus-Time Curve Attained by Time T (%AUC[0-T])
Description: Blood samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); and every 5 mins (from 15 to 30 mins) after each injection. The percent coefficient of variation (CV%) was calculated as 100*(standard deviation/mean). The intra-participant CV% was calculated directly from the 2 replications of each treatment. The CV% for percentage of total AUC is reported from 0 to 30 minutes.
Time Frame: predose up to 30 minutes postdose
Population: Participants who completed all study visits and had evaluable %AUC(0-t) data.
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variance
Groups:
- Insulin Lispro + rHuPH20: Two, subcutaneous (SC) injections of 0.15 units per kilogram (U/kg) insulin lispro with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20), 9 to 42 days apart
- Regular Human Insulin + rHuPH20: Two, subcutaneous (SC) injections of 0.15 units per kilogram (U/kg) regular human insulin (RHI) with 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase (rHuPH20), 9 to 42 days apart
- Insulin Lispro Alone: Two, subcutaneous (SC) injections of 0.15 units per kilogram (U/kg) insulin lispro alone, 9 to 42 days apart
Arm/Group | Insulin Lispro + rHuPH20 | Regular Human Insulin + rHuPH20 | Insulin Lispro Alone
Number analyzed (Participants) | 20 | 20 | 20
percentage of coefficient of variance | 14.04 (11.12) | 23.81 (12.43) | 40.51 (24.30)
Statistical Analysis 1: Comparison: Insulin Lispro + rHuPH20 vs Insulin Lispro Alone; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Treatment comparison for %AUC(0-30). Statistical testing was considered exploratory, with no adjustment for inflation of Type 1 error due to multiplicity of testing; Analysis performed using mixed model with fixed effect for treatment. A compound symmetry covariance matrix among repeated measurements was assumed; LS Mean Difference = 26.47, 90% CI 2-sided [18.22 to 34.71]
Statistical Analysis 2: Comparison: Regular Human Insulin + rHuPH20 vs Insulin Lispro Alone; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 16.70, 90% CI 2-sided [8.45 to 24.94]

2. Secondary Outcome: Time to Early and Late 50% Maximum Serum Insulin Concentration (t[50%Max])
Description: Blood samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); every 30 mins (from 90 to 240 mins); and every 60 mins (from 240 to 480 mins) after each injection.
Time Frame: predose up to 480 minutes postdose
Population: Participants who completed all study visits and had evaluable t(50%max) data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Insulin Lispro + rHuPH20 | Regular Human Insulin + rHuPH20 | Insulin Lispro Alone
Number analyzed (Participants) | 20 | 20 | 20
minutes
  early t(50%max) | 14.14 (3.01) | 21.52 (4.95) | 24.73 (5.16)
  late t(50%max) | 88.14 (16.96) | 136.67 (27.16) | 144.43 (31.79)

3. Secondary Outcome: Peak Serum Insulin Concentration (Cmax)
Description: Cmax was determined as the maximum of all valid serum insulin concentration measurements for each measurement series. Blood samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); every 30 mins (from 90 to 240 mins); and every 60 mins (from 240 to 480 mins) after each injection.
Time Frame: predose up to 480 minutes postdose
Population: Participants who completed all study visits and had evaluable Cmax data.
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | Insulin Lispro + rHuPH20 | Regular Human Insulin + rHuPH20 | Insulin Lispro Alone
Number analyzed (Participants) | 20 | 20 | 20
picomoles per liter (pmol/L) | 782.85 (199.84) | 561.93 (141.88) | 482.40 (119.50)

4. Secondary Outcome: Time to Percentage of Total Glucose Infused
Description: Blood samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); every 30 mins (from 90 to 240 mins); and every 60 mins (from 240 to 480 mins) after each injection. Time to 25%, 50%, and 75% of total glucose infused are summarized.
Time Frame: predose up to 480 minutes postdose
Population: Participants who completed all study visits and had evaluable glucose infusion data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Insulin Lispro + rHuPH20 | Regular Human Insulin + rHuPH20 | Insulin Lispro Alone
Number analyzed (Participants) | 20 | 20 | 20
minutes
  25% | 72.38 (12.50) | 91.58 (15.85) | 99.13 (19.26)
  50% | 118.95 (22.93) | 142.55 (21.31) | 156.83 (30.36)
  75% | 179.23 (40.73) | 203.15 (31.12) | 222.48 (44.44)

5. Secondary Outcome: Percentage of Total Glucose Infused
Description: Blood samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); and every 30 mins (from 90 to 240 mins) after each injection. Percentage of total glucose infused from 0 to 4 hours is summarized.
Time Frame: predose up to 240 minutes postdose
Population: Participants who completed all study visits and had evaluable glucose infusion data.
Measure: Mean (Standard Deviation); unit: percentage of total glucose infused
Arm/Group | Insulin Lispro + rHuPH20 | Regular Human Insulin + rHuPH20 | Insulin Lispro Alone
Number analyzed (Participants) | 20 | 20 | 20
percentage of total glucose infused | 88.70 (9.04) | 85.17 (7.89) | 79.81 (11.27)

6. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) Related to Study Drug
Description: The number of TEAEs related to study drug (as determined by the Investigator) are summarized. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: first dose through 7 to 10 days after last dose
Population: Participants who received at least one dose of study drug (insulin lispro, regular human insulin, or recombinant human hyaluronidase [rHuPH20]).
Measure: Number; unit: events
Arm/Group | Insulin Lispro + rHuPH20 | Regular Human Insulin + rHuPH20 | Insulin Lispro Alone
Number analyzed (Participants) | 22 | 20 | 21
events | 1 | 0 | 3

ADVERSE EVENTS:
Arm/Group | Insulin Lispro + rHuPH20 | Regular Human Insulin + rHuPH20 | Insulin Lispro Alone
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 4/22 | 4/20 | 9/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro + rHuPH20 (N=22) | Regular Human Insulin + rHuPH20 (N=20) | Insulin Lispro Alone (N=21)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 2 (2) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) — A single adverse event of fatigue was undeterminable and could not be assigned to a treatment group due to an incomplete onset date.
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (3)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.